CLINICAL TRIAL: NCT01195246
Title: An Open-Label, Randomized, Multi-Center Study Comparing the Safety and Immunogenicity of HEPLISAV™ to Engerix-B® and Fendrix® in Adults on Hemodialysis Who Have Previously Received Hepatitis B Vaccination and Are Not Seroprotected
Brief Title: Safety and Immunogenicity of HEPLISAV™ a Hepatitis B Virus Vaccine in Adults on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dynavax Technologies Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DV2-HBV-18; 2010-019633-10 (EudraCT Number)
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal failure; renal failure; kidney failure; kidney failure, chronic; chronic kidney failure; hepatitis B virus (HBV) vaccine; hepatitis B vaccine; hepatitis B; hepatitis; HBV; prevention and control; dialysis
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Renal Insufficiency; Hepatitis B; Hepatitis | interventions — Hepatitis B Vaccines; Engerix-B; Fendrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- HEPLISAV (Experimental): 0.5 mL HEPLISAV
  Interventions: Biological: HEPLISAV
- Engerix-B (Active Comparator): 2.0 mL Engerix-B
  Interventions: Biological: Engerix-B
- Fendrix (Active Comparator): 0.5 mL Fendrix
  Interventions: Biological: Fendrix

INTERVENTIONS:
Biological: HEPLISAV — Intramuscular (IM) injection on Day1
  Other Names: Hepatitis B Vaccine (Recombinant), Adjuvanted
  Arms: HEPLISAV
Biological: Engerix-B — Intramuscular (IM) injection on Day 1
  Other Names: Hepatitis B Vaccine (Recombinant)
  Arms: Engerix-B
Biological: Fendrix — Intramuscular (IM) injection on Day 1
  Other Names: Hepatitis B Vaccine (Recombinant)
  Arms: Fendrix

SUMMARY:
The purpose of this study is to compare the immune response to HEPLISAV™ booster injection with the immune response to Engerix-B® and Fendrix® booster vaccinations among patients with end stage renal disease (ESRD) on hemodialysis.

DETAILED DESCRIPTION:
The immune response of HEPLISAV compared with Engerix-B and Fendrix and measured by seroprotection rate (SPR) at 4 weeks after the booster injection

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Has loss of renal function and is receiving hemodialysis treatments
* Is not seroprotected against hepatitis B (has anti-HBs < 10 mIU/mL)
* In the opinion of the investigator, is clinically stable
* Be serum negative for HBsAg, anti-hepatitis B core antigen (HBc), hepatitis C virus (HCV), and HIV
* Is not scheduled to undergo a kidney transplant during the study period
* If female, and of childbearing potential, subject must be: surgically sterile or neither pregnant nor breast-feeding, consistently using a highly effective method of birth control for at least one month prior to study entry, and agrees to use two forms of birth control consistently throughout the study.

Exclusion Criteria:

* If female, is pregnant, breastfeeding, or planning a pregnancy;
* Has a history of or is at high risk for recent exposure to HBV, HCV, or HIV;
* Has known history of autoimmune disease;
* Has history of sensitivity to any component of study vaccines;
* Has a current condition other than renal disease or has substance or alcohol abuse that would interfere with compliance or with interpretation of the study results;
* Is undergoing chemotherapy or expected to receive chemotherapy during the study period; has a diagnosis of cancer within the last 5 years other than squamous or basal cell carcinoma of the skin;
* Has uncontrolled diabetes;
* Has received a kidney transplant previously that is still functioning and requires anti-rejection medication;
* Has received any blood products or immunoglobulin within 3 months prior to study entry, or likely to require infusion of blood products during the study period;
* Has received the following prior to the study injection: 3 days: intravenous iron; 21 days: any inactivated virus or bacterial vaccine; 28 days: any live virus or bacterial vaccine; systemic corticosteroids (more than 3 consecutive days) or other immunomodulators or immune suppressive medication, with the exception of inhaled steroids; granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF); any other investigational medicinal agent;
* At any time: an injection of deoxyribonucleic acid (DNA) plasmids or oligonucleotides; investigational or intradermal hepatitis B vaccine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with seroprotection rate (SPR), defined as the percentage of subjects with anti-HBsAg serum concentration of 10 milli-international unit (mIU)/mL or higher, measured at Week 4 | week 4

SECONDARY OUTCOMES:
Overall incidence of post-injection reactions and adverse events in each treatment group | week 12

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (19):
  - Aschaffenburg
  - Bamberg
  - Berlin
  - Cologne
  - Dresden
  - Düsseldorf
  - Essen
  - Halle
  - Hamburg
  - Hanover
  - Leipzig
  - Madgeburg
  - Mainz
  - Mannheim-Kafertal
  - München
  - Oberschleißheim
  - Rostock
  - Trier
  - Velbert

IPD SHARING:
Plan to Share IPD: Undecided
a/o August 2016, decision is still pending.

REFERENCES:
- See also: Related Info — http://www.dynavax.com